CLINICAL TRIAL: NCT05909956
Title: Effects of Therapeutic Tapping on Clinical Symptoms in Students With Primary Dysmenorrhea
Brief Title: Effects of Therapeutic Tapping in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Sidra Malik
Record Dates: First submitted 2023-06-11; First posted 2023-06-18 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Primary Dysmenorrhea
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KT Group (Experimental): This group will receive Abdominal KT tape (From initial 4 h to 72 h of menstruation). General physio session will also be given to this group.
  Interventions: Other: KinesioTape
- ST Group (Sham Comparator): This group will receive Abdominal KT tape (without strech) from initial 4 h to 72 h of menstruation. General physio session will also be given to this group.
  Interventions: Other: Sham Tape
- CT Group (Other): this group will receive General physical therapy session including Hot pack (3-5min) and General body stretching(stretching of neck & upper trapezius, arm & shoulder girdle, triceps brachii, teres major & minor, quadriceps muscle iliopsoas muscle, adductors muscle, hamstrings muscle) 30-45 sec each, for 7-10 min, (0-4 week) ,45-60sec each, for 10-15 min(4-8week), 15-20 min(8-12week) will be repeated 2 times/day.
  Interventions: Other: General Physio session

INTERVENTIONS:
Other: KinesioTape — The kinesio tape technique, one of the physiotherapy techniques, is an elastic thin band, water-resistant, air-permeable framework to stimulate muscle movements, assist weak muscles (fascia and soft tissue), reduce discomfort and muscle cramps, facilitate proprioceptive input, boost lymph and blood flow, and relieve pain. Participants in the KT group will receive therapeutic tape on the sacral and suprapubic regions with the Star shape and ligament technique (From initial 4 h to 72 h of the menstruation cycle)
  Arms: KT Group
Other: Sham Tape — This group will receive KT tapping without stretch on the sacral and suprapubic region.
  Arms: ST Group
Other: General Physio session — General physical therapy session including Hot pack (3-5min) and General body stretching(stretching of neck & upper trapezius, arm & shoulder girdle, triceps brachii, teres major & minor, quadriceps muscle iliopsoas muscle, adductors muscle, hamstrings muscle) 30-45 sec each, for 7-10 min, (0-4 week) ,45-60sec each, for 10-15 min(4-8week), 15-20 min(8-12week) will be repeated 2 times/day.
  Arms: CT Group

SUMMARY:
Dysmenorrhea is more common among women of reproductive age, as it affects their quality of life and limit their daily activities and normal functioning. The estimates of dysmenorrhea from research conducted all around the world varied widely, from 20% to 90%. This study is planned to determine the effects of KT on clinical symptoms, QOL and academic performance of students with Primary dysmenorrhea.

DETAILED DESCRIPTION:
Literature suggested that kinesio tape technique, one of the effective physiotherapy technique, used for Primary dysmenorrhea, to stimulate muscle movements, assist weak muscles (fascia and soft tissue), reduce discomfort and muscle cramps, facilitate proprioceptive input, boost lymph and blood flow, and relieve pain. This will be a randomized controlled trial, with three groups.

Participants in the experimental group will receive therapeutic tape on the sacral and suprapubic regions with the Star shape and ligament with general physical therapy session. Sham group (ST) group will receive sham taping with general physical therapy session. Participants in Control group (CG) will receive only general physical therapy session.

All groups will be assessed at baseline, at 8th week and 12th week for clinical symptoms, QOL and academic performance.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women with Primary dysmenorrhea
* Aged between 18 and 25 years.
* Having a regular menstruation cycle (28 ± 7 days)
* Severity of menstrual pain on VAS: 4 and over in the previous 6 months.

Exclusion Criteria:

* Secondary dysmenorrhea
* Childbirth, pelvic surgery, use of an intrauterine device,
* Malignant condition
* Chronic medication; antidepressants or oral contraceptives for at least 6 months prior to study
* Not volunteering to participate in the study
* Having an allergy to K.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Changes from Baseline to 8th week
  It is a numeric rating scale from 0 to 10 where 0 represents "no pain" and 10 represents the "worst possible pain.it is used to rate the pain intensity in patients with primary dysmenorrhea.
Visual Analog Scale | Changes from 8th week to 12th week
  It is a numeric rating scale from 0 to 10 where 0 represents "no pain" and 10 represents the "worst possible pain.it is used to rate the pain intensity in patients with primary dysmenorrhea.
Menstrual Symptom Questionnaire | Changes from Baseline to 8th week
  The Menstrual Symptom Questionnaire, a psychometric test, underwent a correlational analysis to determine test-retest reliability. All the items had reliability coefficients equal to or greater than 0.648, and the average coefficient based on Z-score transformation 0.78. It will be used to measure the severity of dysmenorrhea symptoms.
Menstrual Symptom Questionnaire | Changes from 8th week to 12th week
  The Menstrual Symptom Questionnaire, a psychometric test, underwent a correlational analysis to determine test-retest reliability. All the items had reliability coefficients equal to or greater than 0.648, and the average coefficient based on Z-score transformation 0.78. It will be used to measure the severity of dysmenorrhea symptoms.
Health-related life quality | Changes from Baseline to 8th week
  Health-related life quality using the Short Form-36 will be used to measure the pre-post quality of life of the participants and it's a valid and reliable tool used in majority of researches to measure the quality of life.
Health-related life quality | Changes from 8th week to 12th week
  Health-related life quality using the Short Form-36 will be used to measure the pre-post quality of life of the participants and it's a valid and reliable tool used in majority of researches to measure the quality of life.

SECONDARY OUTCOMES:
Self-Structured 20-items Academic Performance questionnaire | Changes from Baseline to 8th week
  It is a 20 items questionnaire, divided under 5 subheadings, in a form of check list "yes or No" response, was developed to measure the impacts of menstrual symptoms on academic performance.
Self-Structured 20-items Academic Performance questionnaire | Changes from 8th week to 12th week
  It is a 20 items questionnaire, divided under 5 subheadings, in a form of check list "yes or No" response, was developed to measure the impacts of menstrual symptoms on academic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Iman girl hostels, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogan H, Eroglu S, Akbayrak T. The effect of kinesio taping and lifestyle changes on pain, body awareness and quality of life in primary dysmenorrhea. Complement Ther Clin Pract. 2020 May;39:101120. doi: 10.1016/j.ctcp.2020.101120. Epub 2020 Feb 22. PMID 32379659
- [Background] Raju J, Suguna M. A study to assess the effect of menstrual symptoms on academic performance among nursing students at selected colleges in Tamil Nadu, India. Int J Appl Res. 2017;3(3):78-80.
- [Background] Mejias-Gil E, Garrido-Ardila EM, Montanero-Fernandez J, Jimenez-Palomares M, Rodriguez-Mansilla J, Gonzalez Lopez-Arza MV. Kinesio Taping vs. Auricular Acupressure for the Personalised Treatment of Primary Dysmenorrhoea: A Pilot Randomized Controlled Trial. J Pers Med. 2021 Aug 19;11(8):809. doi: 10.3390/jpm11080809. PMID 34442453
- [Background] Toprak Celenay S, Kavalci B, Karakus A, Alkan A. Effects of kinesio tape application on pain, anxiety, and menstrual complaints in women with primary dysmenorrhea: A randomized sham-controlled trial. Complement Ther Clin Pract. 2020 May;39:101148. doi: 10.1016/j.ctcp.2020.101148. Epub 2020 Mar 18. PMID 32379680